CLINICAL TRIAL: NCT04324840
Title: A Phase 1b, Open-label, Dose-Finding Study of CC-90010 in Combination With Temozolomide With or Without Radiation Therapy in Subjects With Newly Diagnosed Glioblastoma
Brief Title: A Study of CC-90010 in Combination With Temozolomide With or Without Radiation Therapy in Participants With Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90010-GBM-002; U1111-1248-0496 (Other: WHO); 2019-004122-25 (EudraCT Number)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma
Keywords: CC-90010; Temozolomide; Glioblastoma; NEWLY DIAGNOSED; Radiation therapy; Safety; Tolerability; MTD and RP2D
MeSH Terms: conditions — Glioblastoma; Metatropic dwarfism | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental)
  Interventions: Drug: CC-90010; Drug: Temozolomide; Radiation: Radiotherapy
- Part B - CC-90010 + Temozolomide (TMZ) + Radiotherapy (RT) (Experimental)
  Interventions: Drug: CC-90010; Drug: Temozolomide; Radiation: Radiotherapy
- Part B - Standard TMZ + RT (Other): Control
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: CC-90010 — Specified dose on specified days
  Arms: Part A; Part B - CC-90010 + Temozolomide (TMZ) + Radiotherapy (RT)
Drug: Temozolomide — Specified dose on specified days
  Arms: Part A; Part B - CC-90010 + Temozolomide (TMZ) + Radiotherapy (RT)
Radiation: Radiotherapy — Specified dose on specified days

SUMMARY:
The purpose of this study is to determine the safety and tolerability of CC-90010 when combined with standard of care treatment, temozolomide (TMZ) with or without radiotherapy (RT) in the newly diagnosed WHO Grade IV glioblastoma (ndGBM).

ELIGIBILITY:
Inclusion Criteria:

* Primary isocitrate dehydrogenase (IDH)-wild type newly diagnosed World Health Organization (WHO) Grade IV Glioblastoma
* O6-methylguanine-DNA methyltransferase (MGMT) promoter methylation status must be available prior to randomization
* Karnofsky performance status of ≥70

Exclusion Criteria:

* Indeterminate MGMT promoter methylation status
* Biopsy only of glioblastoma (GBM) at surgery, defined as < 20% resection of enhancing tumor
* Any known metastatic extracranial or leptomeningeal disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to 3 years
  Parts A and B
Incidence of serious adverse events (SAEs) using the NCI CTCAE v5.0 | Up to 3 years
  Parts A and B
Incidence of dose-limiting toxicities (DLTs) | Up to 3 years
  Part A
Maximum Tolerated Dose (MTD) of CC-90010 in combination with Temozolomide (TMZ) | Up to 3 years
  Part A
MTD of CC-90010 in combination with TMZ and Radiation Therapy (RT) | Up to 3 years
  Part A
Recommended Phase 2 Dose (RP2D) of CC-90010 in combination with TMZ | Up to 3 years
  Part A
RP2D of CC-90010 in combination with TMZ and RT | Up to 3 years
  Part A
Median Progression-free survival (PFS) in Arm A vs Arm B | Up to 12 months
  Part B
Hazard ratio for PFS in Arm A vs Arm B | Up to 12 months
  Part B

SECONDARY OUTCOMES:
Progression-free survival (PFS) defined as the time from the first dose of CC-90010 to the first occurrence of disease progression or death from any cause | Up to 5 years
  Parts A and B
Overall survival (OS) measured as the time from the first dose of CC-90010 to death due to any cause and will be analyzed in a manner similar to that described for PFS | Up to 5 years
  Parts A and B
Duration of therapy (DoT) in Arm A vs Arm B | Up to 5 years
  Part B
Response by Response Assessment in Neuro-Oncology (RANO) criteria | Up to 5 years
  Parts A and B
Pharmacokinetics - Maximum observed plasma concentration (Cmax) | Up to 2 years
  Parts A and B
Pharmacokinetics - Area under the plasma concentration time-curve (AUC) | Up to 2 years
  Parts A and B
Pharmacokinetics - Time to maximum plasma concentration (Tmax) | Up to 2 years
  Parts A and B

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- Local Institution - 800, New York, New York, United States
- Denmark (3):
  - Local Institution - 503, Aalborg
  - Local Institution - 501, Copenhagen
  - Local Institution - 500, Odense
- Italy (4):
  - Local Institution - 202, Milan
  - Local Institution - 201, Milan
  - Local Institution - 204, Padua
  - Local Institution - 200, Verona
- Netherlands (4):
  - Local Institution - 408, Leiden, South Holland
  - Local Institution - 405, Amsterdam
  - Local Institution - 400, Rotterdam
  - Local Institution - 401, Utrecht
- Local Institution - 600, Oslo, Norway
- Spain (12):
  - Local Institution - 311, A Coruña
  - Local Institution - 306, Barcelona
  - Local Institution - 302, Barcelona
  - Local Institution - 303, Barcelona
  - Local Institution - 307, Hospitalet de Llobregat, Barcelona
  - Local Institution - 304, Madrid
  - Local Institution - 301, Madrid
  - Local Institution - 300, Madrid
  - Local Institution - 310, Pamplona
  - Local Institution - 309, Seville
  - Local Institution - 305, Valencia
  - Local Institution - 312, Vigo
- Sweden (4):
  - Local Institution - 702, Gothenburg
  - Local Institution - 701, Lund
  - Local Institution - 700, Solna
  - Local Institution - 703, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Moreno V, Manuel Sepulveda J, Reardon DA, Perez-Nunez A, Gonzalez Leon P, Hanna B, Filvaroff E, Aronchik I, Chang H, Amoroso B, Zuraek M, Sanchez-Perez T, Mendez C, Stephens D, Nikolova Z, Vogelbaum MA. Trotabresib, an oral potent bromodomain and extraterminal inhibitor, in patients with high-grade gliomas: A phase I, "window-of-opportunity" study. Neuro Oncol. 2023 Jun 2;25(6):1113-1122. doi: 10.1093/neuonc/noac263. PMID 36455228
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04324840.html